CLINICAL TRIAL: NCT02954692
Title: A National, Multicenter, Prospective, Interventional, Open-label, Single-arm, 24-Week Phase IV Study to Evaluate the Effectiveness and Safety of Initiation and Titration of Insulin Glargine U300 in Insulin-naïve Patients With T2DM Inadequately Controlled on OAD Treatment in Turkey
Brief Title: A Study to Evaluate the Effectiveness and Safety Initiation and Titration of Insulin Glargine (U300) in Insulin-naïve Patients With Type 2 Diabetes Mellitus (T2DM) Controlled on Oral Antidiabetic Drug Treatment in Turkey
Acronym: EASE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLARGL07921; U1111-1183-8755 (Other: UTN)
Record Dates: First submitted 2016-11-02; First posted 2016-11-03 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Metformin; Sulfonylurea Compounds; meglitinide; Thiazolidinediones; Glycoside Hydrolase Inhibitors; Dipeptidyl Peptidase 4; Sodium-Glucose Transporter 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin glargine (U300) (Experimental): Insulin glargine (U300) will be administered daily through subcutaneous injection, and thereafter, dose will be titrated weekly (preferably 3-4 days) as needed. Background non-insulin anti-diabetic drugs approved for use in combination with insulin according to local labelling, will be permitted, with the exception of Thiazolidinediones (TZDs), which must be stopped at the time of basal insulin initiation.
  Interventions: Drug: INSULIN GLARGINE (U300); Drug: metformin; Drug: sulfonylurea; Drug: meglitinides; Drug: thiazolidinediones; Drug: alpha-glucosidase inhibitors; Drug: GLP1 Receptor Agonist; Drug: Dipeptidyl peptidase-IV (DPP-IV) inhibitors; Drug: Sodium-glucose transport-2 (SGLT-2) inhibitors

INTERVENTIONS:
Drug: INSULIN GLARGINE (U300) — Pharmaceutical form: pen for injection
  Route of administration: subcutaneous
  Other Names: HOE901
Drug: metformin — Pharmaceutical form: tablet
  Route of administration: oral
Drug: sulfonylurea — Pharmaceutical form: tablet
  Route of administration: oral
Drug: meglitinides — Pharmaceutical form: tablet
  Route of administration: oral
Drug: thiazolidinediones — Pharmaceutical form: tablet
  Route of administration: oral
Drug: alpha-glucosidase inhibitors — Pharmaceutical form: tablet
  Route of administration: oral
Drug: GLP1 Receptor Agonist — Pharmaceutical form: pen for injection
  Route of administration: subcutaneous
Drug: Dipeptidyl peptidase-IV (DPP-IV) inhibitors — Pharmaceutical form: tablet
  Route of administration: oral
Drug: Sodium-glucose transport-2 (SGLT-2) inhibitors — Pharmaceutical form: tablet
  Route of administration: oral

SUMMARY:
Primary Objective:

To assess the mean change in HbA1c (glycated haemoglobin).

Secondary Objectives:

To evaluate the efficacy and safety of the titration of insulin glargine U300 in terms of:

* Targeted HbA1c;
* Targeted fasting self- monitoring blood glucose (SMBG);
* Hypoglycemic events;
* Adverse events;
* Quality of life assessment by DTSQs (Diabetes Treatment Satisfaction Questionnaire status) and DTSQc (Diabetes Treatment Satisfaction Questionnaire change);
* Blood glucose fluctuation by using continuous glucose monitoring system (CGMS) in subgroup patients.

DETAILED DESCRIPTION:
The total study duration per patient will be 27 weeks (2 weeks of screening, 24 weeks on treatment, and 1 week follow-up period).

ELIGIBILITY:
Inclusion criteria :

* Adult patients with type 2 diabetes mellitus (≥18 years of age).
* Type 2 diabetes mellitus diagnosis ≥1 year.
* Treated with ≥1 oral antidiabetics (±glucagon like peptid-1 (GLP-1) analogue) without insulin, for at least 6 months and HbA1c level between 8-11% (insulin-naïve).
* Stable antidiabetic treatment for at least 3 months.
* Willingness to adherence to treatment and titration (including self-injection, self- monitoring blood glucose [SMBG]).
* Signed informed consent obtained.

Exclusion criteria:

* Age <18 years old.
* Type 1 diabetes mellitus.
* Having secondary type 2 diabetes mellitus.
* Use of any insulin therapy including premix, basal plus/basal bolus regimen from the diagnosis.
* History of hypoglycemia unawareness.
* Known hypersensitivity/intolerance to insulin glargine or any of its excipients.
* Have any condition (including known substance or alcohol abuse or psychiatric disorder) that precludes the patient from following and completing the study protocol.
* Use of systemic glucocorticoids for two weeks or more within 12 weeks prior to the time of screening.
* Pregnant or lactating women.
* Participation in another clinical trial.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2016-11-30; Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in HbA1c | Baseline, Week 24

SECONDARY OUTCOMES:
Percentage of patients achieving targeted fasting self-monitored blood glucose (SMBG) without experiencing severe and/or confirmed hypoglycemia ≤70mg/dL and <54 mg/dL | At Weeks 12 and 24
Percentage of patients reaching targeted fasting SMBG (80-130 mg/dL) | At Weeks 12 and 24
Duration to reach target pre-breakfast SMBG | Baseline, Week 24
Mean change from baseline in HbA1c | Baseline, Week 12
Mean change from baseline in SMBG | Baseline, Weeks 12, and 24
Mean change from baseline in fasting plasma glucose (FPG) | Baseline, Weeks 12, and 24
Mean change from baseline in Diabetes Treatment Satisfaction Questionnaire (DTSO) scores | Baseline, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Turkey, Turkey (Türkiye)